CLINICAL TRIAL: NCT05906953
Title: A Phase 1/2, Open-label, Multi-national, Multiple-cohort, Dose-escalation Study to Evaluate the Safety, Tolerability, and Efficacy of HG004 Gene Therapy in Subjects with RPE65-associated Leber Congenital Amaurosis Type 2 (LCA2)
Brief Title: Safety and Efficacy Trial of HG004 for Leber Congenital Amaurosis Related to Rpe65 Gene Mutations (STAR)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: HuidaGene Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HG00402
Record Dates: First submitted 2023-05-09; First posted 2023-06-18 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Leber Congenital Amaurosis; Inherited Retinal Diseases Caused by RPE65 Mutations
Keywords: IRD; LCA; LCA2
MeSH Terms: conditions — Leber Congenital Amaurosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- HG004 (Experimental)
  Interventions: Drug: HG004

INTERVENTIONS:
Drug: HG004 — Low dose Medium dose High dose

SUMMARY:
The purpose of the study is to determine whether HG004 as gene therapy is safe and effective for the treatment of Leber Congenital Amaurosis caused by mutations in RPE65 gene.

ELIGIBILITY:
Inclusion Criteria:

* Male or females between 6 and 50 years of age at the time of signing the informed consent form.
* Willing to adhere to protocol as evidenced by written informed consent or parental permission and subject assent.
* Clinical confirmed diagnosis of Leber congenital amaurosis (LCA) and molecular diagnosis of LCA due to RPE65 mutations.
* Ability to perform tests of visual and retinal function.
* Visual acuity of ≤ 20/80 or visual field less than 20 degrees in the eye to be injected.
* Acceptable hematology, clinical chemistry, and urine laboratory parameters.

Exclusion Criteria:

* Pre-existing eye conditions that would preclude the planned surgery or interfere with interpretation of study endpoints or complications of surgery (e.g., glaucoma requiring upcoming surgery, corneal or significant lenticular opacities).
* Presence of epiretinal membrane by OCT.
* Complicating systemic diseases or clinically significant abnormal baseline laboratory values.
* Complicating systemic diseases would include those in which the disease itself, or the treatment for the disease, can alter ocular function.
* Prior ocular surgery within six months.
* Prior gene therapy or oligonucleotide therapy treatments.
* Any condition which leads the investigator to believe that the participant cannot comply with the protocol requirements or that may place the participant at an unacceptable risk for participation.

Ages: 6 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of ocular and non-ocular adverse events | 52 weeks

SECONDARY OUTCOMES:
Change from baseline in Best Corrected Visual Acuity (BCVA) of letters based on the Early Treatment Diabetic Retionpathy Study (ETDRS) chart | 52 weeks
Change from baseline in visual fields of full-field stimulus threshold test in log cd.s/m2. | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — HuidaGene Therapeutics Co., Ltd.
Locations (3):
- United States (2):
  - Research Site, Sacramento, California
  - Research Site, Houston, Texas
- Research Site, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No